CLINICAL TRIAL: NCT02019212
Title: Prognostic Value of Stress SPECT Myocardial Perfusion Imaging With Half Dose 99mTc-tetrofosmin
Status: Completed | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Renee Hessian, MD, Ottawa Heart Institute Research Corporation
Other Study IDs: 20130446-01H
Record Dates: First submitted 2013-10-09; First posted 2013-12-24 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Disease
Keywords: 99mTc-tetrofosmin; myocardial perfusion imaging; SPECT; radiation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MPI Perfusion Imaging: Clinical patients who have undergone myocardial perfusion imaging with 99mTc

SUMMARY:
The purpose of this study is to evaluate the quality and prognostic ability of low dose 99mTc-tetrofosmin Myocardial Perfusion SPECT Imaging.

DETAILED DESCRIPTION:
The objective of this study is to determine if myocardial perfusion imaging (MPI) using a new SPECT reconstruction software and a low dose (LD) of 99mTC-tetrofosmin will provide equal quality and prognostic value as a full dose (FD) of 99mTc-tetrofosmin myocardial perfusion SPECT imaging methodology.

The images of clinical patients from the Diagnostic Imaging Department will be assessed and compared for image quality and myocardial perfusion. The outcomes of participants that have had FD studies will be compared to those who have had LD studies. Consented participants will be contacted and will be asked to provide information on their cardiovascular health since the date of their LD or FD scan, such as non fatal myocardial infarction, death, congestive heart failure, admission to hospital with chest pain, further cardiac diagnostic testing, including angiography and early and late revascularization. The event information will be tabulated at 6, 12, 18, and 24 months for the LD and FD studies.

The study hypothesizes that there will be no difference in the quality and prognostic value between the LD and FD 99mTc-tetrofosmin SPECT MPI imaging protocols. The study hypothesizes that there will be no increase in repeat diagnostic testing and angiography with using the LD imaging protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have completed the FD and LD MPI studies on the GE Infinia Haweye or GE NM 530 (CZT crystal) cameras
* Retrospective participants must consent to the study interview(s) for data collection
* Prospective participants must consent to follow up for data collection

Exclusion Criteria:

* Unwilling to consent to data collection either retrospectively or in follow up prospectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical patients who have undergone myocardial perfusion imaging.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-10-27 (Actual); Study Completion 2016-10-27 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Outcomes | 15 minutes
  The primary objective is to compare the cardiovascular outcomes of participants that have had FD studies to those that have had LD studies. These cardiovascular outcomes include myocardial infarction, death, congestive heart failure, hospitalization with chest pain, further diagnostic testing, including angioplasty, and early and late revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Renée Hessian, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Insitute, Ottawa, Ontario, Canada